CLINICAL TRIAL: NCT00909194
Title: Juvenile Primary Fibromyalgia in a Female Adolescent Psychiatric Population
Brief Title: Juvenile Primary Fibromyalgia Syndrome (JPFS) in an Adolescent Psychiatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joel Thompson (Other)
Responsible Party: Sponsor-Investigator, Joel Thompson, Clinical trial compliance administrator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIBRO1
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Juvenile Primary Fibromyalgia Syndrome
Keywords: Juvenile Primary Fibromyalgia; Adolescents; Psychiatry
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Educational Seminar on Juvenile Primary Fibromyalgia Syndrome and CD-guided total body relaxation technique
  Interventions: Behavioral: Psychoeducational Seminar and Relaxation Technique
- Control (No Intervention): Control Arm consisted of an educational seminar on skin care

INTERVENTIONS:
Behavioral: Psychoeducational Seminar and Relaxation Technique — Psychoeducational seminar on Juvenile Primary Fibromyalgia (pain management, diet, exercise and sleep hygiene) followed by a total body relaxation technique
  Arms: Intervention

SUMMARY:
The purpose of this study was to identify clinical characteristics and estimate the prevalence of Juvenile Primary Fibromyalgia in a female inpatient psychiatric population. The secondary purpose of this study was to determine the efficacy of an intervention (psychoeducational seminar and relaxation technique) on reducing the symptoms of Juvenile Primary Fibromyalgia Syndrome. We looked at the short-term and long-term effects of this intervention in comparison to the control (skin care seminar).

DETAILED DESCRIPTION:
The specific aims of phase one of this study were to estimate the prevalence of Juvenile Primary Fibromyalgia Syndrome (JPFS) in an inpatient female psychiatric population and to identify characteristics associated with JPFS in this population. We chose to explore two primary hypotheses. Because of the common link between adult fibromyalgia and anxiety and depression, we hypothesize that those with JPFS will score higher on measures of these symptoms. Given the adult literature on the suspected link between physical and or sexual abuse and adult fibromyalgia, we also hypothesized that adolescents who meet criteria for JPFS will have higher rates of sexual and physical abuse.

The other specific aim of this study was to determine the short- and long-term impact of an intervention on reduction of JPFS symptoms. The intervention was a psychoeducational seminar on JPFS (pain management, diet, exercise and sleep hygiene) followed by a relaxation technique (audio-guided CD). The control group was involved in an educational seminar on skin care (WITHOUT relaxation technique). Study measures were obtained immediately before and after the intervention/control seminars (short-term) and 8 weeks after discharge (long-term). Each group was discharged with a CD player and CD with relaxation technique or skin care seminar. Participants recorded the use of the CD's and completed follow up questionnaires 8 weeks after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to inpatient child psychiatric facility
* Between 12-18 years of age
* in parental or family (relative as guardian) custody

Exclusion Criteria:

* In state custody
* low intellectual functioning (i.e. IQ less than or equal to 70)
* active psychosis

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To characterize adolescents who are admitted to an inpatient psychiatric unit and meet criteria for JPFS

SECONDARY OUTCOMES:
To determine the efficacy of an intervention on functioning and well-being (short-term and long-term) | Immediately after intervention and 8 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Lommel, DO, MHA, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States